CLINICAL TRIAL: NCT06501794
Title: Pilot Study: Use of the Saccadometer to Detect Characteristic Saccadic Peak Velocity in Myasthenia Gravis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UoL001162
Record Dates: First submitted 2016-02-26; First posted 2024-07-15 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-07

CONDITIONS: Myasthenia Gravis
Keywords: Saccades
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Myasthenia Gravis (Other): Participants with a confirmed diagnosis of Myasthenia Gravis
  Interventions: Device: Quantitative measurement of eye movements

INTERVENTIONS:
Device: Quantitative measurement of eye movements — Saccadometer © - diagnostic device: non-invasive quantitative assessment of eye movement

SUMMARY:
Fast eye movements have been shown to demonstrate characteristics that are specific to myasthenia gravis that are not present in other eye movement disorders. It is possible to measure these eye movements and potentially identify these characteristics using new portable eye movement testing equipment. The aim of this pilot study is to discover if these characteristics can be identified using portable eye movement testing equipment in patients with a confirmed diagnosis of myasthenia gravis.

DETAILED DESCRIPTION:
The diagnosis of Myasthenia Gravis (MG) can be challenging, particularly in its ocular manifestation with current clinical procedures. Previous research has shown that fast eye movements in patients suffering with MG have quite specific characteristics that can be used to correctly diagnose the condition. The Saccadometer is a portable eye movement testing device that may provide the ability to detect the characteristics of fast eye movements that Myasthenia patients alone demonstrate - specifically these are hyperfast movements that are present when slower eye movements are impaired by the disease process. These fast movement characteristics are not present in defects of eye movements due to other aetiologies.

Saccadic properties of a small group of patients with a confirmed diagnosis of MG will be measured to identify if characteristic hyperfast saccades are present.

ELIGIBILITY:
Inclusion Criteria:

Patient participants

* Confirmed diagnosis of Myasthenia Gravis by either a positive acetylcholine antibody serum test (AChR) and/or a positive single fibre electromyograph (SFEMG) test.
* Patient participants must have also had at least one episode of diplopia and/or eye movement abnormality attributed to their diagnosis of MG.

Healthy participants:

* Must have no history of eye movement abnormality
* No have no history of other auto-immune disease (specifically diabetes, Thyroid Eye Disease and Chronic External Ophthalmoplegia).

Exclusion Criteria:

* Patients without confirmed Myasthenia Gravis diagnosis by means of either a positive AChR serum test and/or a positive SFEMG test.
* Patients with confirmed Myasthenia Gravis who have not had at least one episode of diplopia and or ptosis.
* Patients with current or previous episodes of ocular motility dysfunction that have a confirmed diagnosis other than Myasthenia Gravis.
* Any healthy participant found to have an abnormality of vision or eye movement upon screening or a history of auto-immune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Saccadic Peak Velocity | Measured at first and only contact point within study i.e. day one and then not tested again
  Participants will be recruited, consented and tested at a single visit during their routine clinical visit, up to one year after being recruited. Quantitative assessment of their eye movements using the Saccadometer will be assessed at that point of contact and the outcome measure recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Murray, MRes, Principal Investigator — University of Liverpool

IPD SHARING:
Plan to Share IPD: No